CLINICAL TRIAL: NCT01373905
Title: Stepwise PEEP Elevation With Determination of the Alveolar Collapsing Pressure Versus Sustained Lung Inflation as a Recruitment Maneuver in Patients With ARDS
Brief Title: Stepwise Positive End Expiratory Pressure Elevation For Lung Recruitment in Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Vice-Dean for Post-Graduate Studies and Research, faculty of Medicine - university of Alexandria
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Faculty of Medicine12.12.2006
Record Dates: First submitted 2011-06-08; First posted 2011-06-15 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2008-02

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; PEEP; Recruitment maneuver
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sustained lung inflation (Active Comparator): recruitment was done using CPAP of 30 Cm/ H2o for 30 seconds
  Interventions: Procedure: Recruitment maneuver
- Stepwise PEEP elevation (Active Comparator): Recruitment was done using stepwise elevation of PEEP followed by determination of the alveolar collapsing pressure
  Interventions: Procedure: Recruitment maneuver

INTERVENTIONS:
Procedure: Recruitment maneuver — group I: Recruitment by CPAP 30 cm/H2o for 30 seconds group II: Using pressure controlled ventilation with end-inspiratory minus end-expiratory pressure of 15 cmH2O, respiratory rate of 10-15 C / min. PEEP was increased by 5 cm/ H2O every 2 minutes till Maximum of 40 cmH2O, patient was considered recruited if PaO2 of 250 mmHg was achieved. Then progressive decreases of PEEP in steps of 2 cmH2O every 2 minutes till PaO2 dropped by a 10% or more (alveolar collapsing pressure)
Procedure: recruitment maneuver — recruitment as done by CPAP 30 cm/ H2o for 30 seconds or by stepwise elevation of PEEP by 5 cm/ H20 till 40 Cm/ H2o

SUMMARY:
Acute respiratory distress syndrome is a severe lung disease caused by a variety of direct and indirect issues. It is characterized by inflammation of the lung parenchyma leading to impaired gas exchange and persistent hypoxemia. This condition is often fatal, usually requiring mechanical ventilation. Recruitment maneuver aimed to enhance the effect of mechanical ventilation.The objective of this study was to compare safety and efficacy of two lung recruitment maneuvers.

DETAILED DESCRIPTION:
In patients with acute respiratory distress syndrome (ARDS), protective lung strategy and positive end expiratory pressure (PEEP) therapy should be started as early as possible to avoid lung damage by high pressures, volumes and fraction of inspired oxygen (FiO2). Recruitment is a strategy aiming at re-expanding the collapsed lung tissue and then maintaining an adequate level of PEEP to prevent subsequent de-recruitment. The objective of this study was to compare safety and efficacy of two lung recruitment maneuvers (RM): stepwise PEEP elevation with determination of the alveolar collapsing pressure versus sustained lung inflation in ARDS patients

ELIGIBILITY:
Inclusion Criteria:

* ARDS
* lung injury score more than 2.5
* on mechanical ventilation

Exclusion Criteria:

* hemodynamic instability
* left heart failure
* pneumothorax
* COPD
* restrictive lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 30 days

SECONDARY OUTCOMES:
Efficacy | 24 hours
  oxygenation index, compliance and lung infiltration

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M El-Mehalawy, MD, Principal Investigator — Faculty of Medicine, Alexandria University, Egypt
Locations (1):
- Faculty of Medicine, Alexandria, Alexandria Governorate, Egypt

REFERENCES:
- [Background] Borges JB, Okamoto VN, Matos GF, Caramez MP, Arantes PR, Barros F, Souza CE, Victorino JA, Kacmarek RM, Barbas CS, Carvalho CR, Amato MB. Reversibility of lung collapse and hypoxemia in early acute respiratory distress syndrome. Am J Respir Crit Care Med. 2006 Aug 1;174(3):268-78. doi: 10.1164/rccm.200506-976OC. Epub 2006 May 11. PMID 16690982